CLINICAL TRIAL: NCT01826344
Title: The Vascutek Custom Fenestrated Anaconda Post-Market Surveillance Study
Status: Terminated | Type: Observational
Sponsor: Vascutek Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CFD001
Record Dates: First submitted 2013-04-03; First posted 2013-04-08 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Abdominal Aortic Aneurysms (AAA)
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multicentre, prospective, observational post-market registry (follow-up 1 month, 1 year, 2 years, 3 years, 4 years and 5 years) to monitor the post-market clinical safety and effectiveness of the Vascutek AnacondaTM Custom Fenestrated Stent Graft in patients with a short infrarenal neck of <15mm or juxta-renal abdominal aortic aneurysms who, in the opinion of the treating physician, are anatomically suitable for the AnacondaTM Custom Fenestrated Stent Graft and for whom a customised medical device is required.

DETAILED DESCRIPTION:
AnacondaTM Custom Fenestrated Devices (CFD) are designed for the endovascular repair of abdominal aortic aneurysms (AAA) for cases where the aneurysm extends superiorly very close to or involving the renal arteries, leaving insufficient neck length for infrarenal device sealing. The non-CE marked devices are custom designed based on CT scan data of the patient's aorta and regulated in accordance with the Medical Device Directive (93/42/EEC) and associated country specific regulations as applicable.

The proximal end of the AnacondaTM fenestrated body device is positioned suprarenally, where it seals and fixates in the vessel by means of rings comprised of multiple turns of fine nitinol wire, attached to the fabric with polyester sutures, creating a self-expanding stent which provides a conformable seal with the vessel wall and assists in anchoring of the device. Nitinol hooks provide secure fixation within the suprarenal aorta. The saddle shape of the rings allows the superior mesenteric artery (SMA) or celiac artery to be accommodated in the valley of the top ring saddle in some cases.

The objective of the registry is to provide long term (5 year) safety and effectiveness data of all patients who consent to their data to be used in the registry. This data aims to demonstrate that the Vascutek AnacondaTM Custom Fenestrated Stent Graft is safe and effective in patients with a short infrarenal neck of <15mm or juxta-renal abdominal aortic aneurysms who, in the opinion of the treating physician, are anatomically suitable for the AnacondaTM Custom Fenestrated Stent Graft.

ELIGIBILITY:
Inclusion Criteria:

A patient with juxta renal abdominal aortic aneurysms (AAA) who, in the opinion of the treating physician, is anatomically suitable for the Anaconda Fenestrated Graft and for whom a customised medical device is required.

Exclusion Criteria:

1. Ruptured or symptomatic aneurysm
2. Clinically significant concomitant medical disease or infection
3. Connective Tissue Disease (e.g. Marfan's Syndrome)
4. Known allergy to nitinol, polyester or contrast medium
5. Excessive tortuosity of access vessels (femoral or iliac arteries)
6. Landing zone of less than 10mm in the visceral segment of the aorta
7. Inability to comply to follow up protocol
8. Access vessels less than 6mm in diameter
9. Diseased or excessively tortuous access to target vessels
10. Target vessels of less than 5mm in calibre
11. Excessive calcification or thrombus at the intended landing zone which could affect sealing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a short infrarenal neck of <15mm or juxta-renal abdominal aortic aneurysms who, in the opinion of the treating physician, are anatomically suitable for the AnacondaTM Custom Fenestrated Stent Graft and for whom a customised medical device is required.
Sampling Method: Non-Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2010-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To monitor the the post-market clinical safety and effectiveness of the Vascutek AnacondaTM Custom Fenestrated Stent Graft | For 5 years post-implant
  To monitor the post-market clinical safety and effectiveness of the Vascutek AnacondaTM Custom Fenestrated Stent Graft in patients with a short infrarenal neck of <15mm or juxta-renal abdominal aortic aneurysms who, in the opinion of the treating physician, are anatomically suitable for the AnacondaTM Custom Fenestrated Stent Graft and for whom a customised medical device is required.

CONTACTS AND LOCATIONS:
Locations (71):
- Austria (2):
  - Kaiser Franz Josef Spital, Vienna
  - Krankenhaus Hietzing, Vienna
- Belgium (5):
  - Imelda Hospital, Bonheiden
  - St Luc Brussels, Brussels
  - University Hospital, Brussels, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - H.-Hartziekenhuis Roeselare-Menen, Roeselare
- Canada (8):
  - Peter Lougheed Centre, Calgary
  - QE2 Hospital, Halifax
  - London Health Sciences Centre, London, Ontario
  - Royal Victoria Hospital, Montreal
  - The Ottawa Hospital, Ottawa
  - St Clare's Mercy Hospital, St. Johns
  - Toronto General Hospital, Toronto
  - Health Science Centre, Winnipeg
- France (7):
  - Hopital Pellegrin, Bordeaux
  - CHU Henri Mondor, Créteil
  - Chirurgien Vasculaire, Draguignan
  - Clinique Ambrose Paré, Nancy
  - La Pitie, Paris
  - Le Plessis Robinson, Paris
  - CHU Tours, Tours
- Germany (20):
  - Luisenhospital - Aachen, Aachen
  - University Hospital Aachen, Aachen
  - Klinikum Augsburg, Augsburg
  - Red Cross hospital clinic, Bremen
  - University of Cologne, Cologne
  - Klinikum Frankfurt Hochst, Frankfurt
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Krankenhaus Freital, Freital
  - Chirurgie am Waldweg, Göttingen
  - University of Groningen, Gröningen
  - Asklepios Klinik Altona, Hamburg
  - Medical Care Centre for Vascular Diseases, Hamm
  - Marienhospital, Kevelaer
  - Bonifacius Hospital, Lingen
  - University Hospital, Munich
  - DRK Krankenhaus Neustrelitz, Neustrelitz
  - Krankenhaus Barmherzige Bruder, Regensburg
  - University Hospital, Regensburg
  - Klinikum Solingen, Solingen
  - Marien-Hospital Witten, Witten
- Italy (4):
  - University of Bologna, Bologna
  - Ospedale San Francesco, Nuoro
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervel, Palermo
  - San Filippo Neri Hospital, Rome
- Centre Cardio Thoracique, Monaco, Monaco
- Netherlands (5):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Medisch Spectrum Twente, Enschede
  - Maastricht University Medical Centre, Maastricht
  - Erasmus University, Rotterdam
  - Isala Klinieken, Zwolle
- Spain (4):
  - Hospital Donostia, Donostia / San Sebastian
  - Hospital Universitario La Paz, Madrid
  - Hospital de Navarra, Pamplona
  - Hospital Universitari Parc Tauli, Sabadell
- Uppsala University, Uppsala, Sweden
- Switzerland (2):
  - University Hospital Bern, Bern
  - Kantonsspital Graubunden, Chur
- United Kingdom (12):
  - Royal Derby Hospital, Derby
  - Frimley Park Hospital, Frimley
  - Western Infirmary/Gartnavel, Glasgow
  - Leeds General Infirmary, Leeds
  - Leicester Royal Infirmary, Leicester
  - Imperial (St Mary's / Charing X) Hospital, London
  - Kings College Hospital, London
  - The Royal Free Hospital, London
  - The Royal London Hospital, London
  - Freeman Hospital, Newcastle
  - John Radcliffe Hospital, Oxford
  - Royal Preston Hospital, Preston